CLINICAL TRIAL: NCT04602871
Title: Early Detection of the 2019 Novel Coronavirus (SARS-CoV-2) Using Breath Analysis - Feasibility Study
Brief Title: Early Detection of COVID-19 Using Breath Analysis - Feasibility Study
Acronym: COVID-19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Scentech Medical Technologies Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Cov-2-2020
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2022-05-10 (Actual); Status verified 2020-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID 19 Positive patients (Experimental): Patients with COVID-19, qPCR for SARS-CoV-2 confirmed
  Interventions: Diagnostic Test: Breath Biopsy
- Healthy subjects (Other): COVID-19 Negative subjects
  Interventions: Diagnostic Test: Breath Biopsy

INTERVENTIONS:
Diagnostic Test: Breath Biopsy — Breath Biopsy sampling using the ReCIVA® Breath Sampler

SUMMARY:
Early Detection of COVID-19 Using Breath Analysis -Feasibility Study.

DETAILED DESCRIPTION:
An interventional diagnostic prospective study study with risks and minimal constraints.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized group:

* Age 18 to 75 years at the time of consent
* Positive results for SARS-CoV-2
* Capable of understanding written and/or spoken language
* Able to provide informed consent
* Was not treated with Anti-viral drugs
* Not a pregnant woman

Healthy group:

* Healthy volunteers
* Age 18 to 75 years at the time of consent
* No history of COVID-19
* Capable of understanding written and/or spoken language
* Able to provide informed consent
* Was not treated with Anti-viral drugs
* Not a pregnant woman

Sexes Eligible for Study: All

Exclusion Criteria:

Hospitalized group:

* Age under 18 years old
* (Anticipated) inability to complete breath sampling procedure due to e.g. hyper- or hypoventilation, respiratory failure or claustrophobia when wearing the sampling mask
* Persons under guardianship or deprived of liberty
* Patients with the following diseases: Cancer, Asthma, Chronic Respiratory Disease

Healthy group:

* Age under 18 years old
* History of COVID-19
* Persons under guardianship or deprived of liberty
* Subjects with the following diseases: Cancer, Asthma, Chronic Respiratory Disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-07-03 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Correlation between Volatile Organic Compounds pattern in-breath biopsy and COVID-19 detection. | Through the study completion, up to 3 months.
  Correlation between Volatile Organic Compounds found in breath biopsy chromatography and COVID-19 detection in a swab test.

SECONDARY OUTCOMES:
Correlation between Volatile Organic Compounds pattern and the course of the disease | Through the study completion, up to 3 months.
  Correlation between Volatile Organic Compounds found in breath biopsy chromatography and COVID-19 detection intensity in a swab test.

CONTACTS AND LOCATIONS:
Overall Officials: David Shitrit, MD, Principal Investigator — Meir Medical Center, Kfar Saba, Israel
Locations (2):
- Israel (2):
  - Soroka Medical Center, Beersheba
  - Meir Medical Center, Kfar Saba

IPD SHARING:
Plan to Share IPD: No
No IPDs are to be shared with other researchers.